CLINICAL TRIAL: NCT00551200
Title: A Phase 2, Open-Label, Switch-Over, Dose-Escalation Study of the Safety and Tolerability of HPN-100 Compared to Buphenyl® (Sodium Phenylbutyrate) in Patients With Urea Cycle Disorders
Brief Title: Dose-Escalation Safety Study of HPN-100 to Treat Urea Cycle Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP1204-003 (HPN-100-003)
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Urea Cycle Disorders
Keywords: Buphenyl; Sodium Phenylbutyrate; Urea Cycle Disorder; UCD
MeSH Terms: conditions — Urea Cycle Disorders, Inborn | interventions — glycerol phenylbutyrate; 4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BUPHENYL® to HPN-100 vs. HPN-100 (Active Comparator): Buphenyl treatment for one week was followed by dose escalation to HPN-100. Dose of Buphenyl was gradually decreased while HPN-100 dose was gradually increased until subject reached dosing of 100% HPN-100. HPN-100 at 100% of the dose was given for 1 week before subject was switched back to original Buphenyl treatment.
  Interventions: Drug: HPN-100; Drug: BUPHENYL®

INTERVENTIONS:
Drug: HPN-100 — Subjects will be taking prescribed dose of Buphenyl® TID (not to exceed 20g/day) at least two weeks prior to enrollment. Subjects will take prescribed dose of Buphenyl® TID for first week of study, and then switch over to HPN-100 TID during a dose-escalation phase. The dose of HPN-100 will be increased and the dose of Buphenyl® will be decreased each week by 50 mg/kg until entire daily dose of phenylbutyrate is HPN-100. Target HPN-100 dose will contain the same amount of phenylbutyrate as the subject's prescribed daily dose of Buphenyl®. Subject will take HPN-100 alone for one week and then switch back to previous dose of Buphenyl for the last week of the study.
Drug: BUPHENYL® — BUPHENYL® (sodium phenylbutyrate) tablets and powder have been approved for marketing in the United States since 1996 as an adjunctive therapy in the long-term management of patients with UCDs involving deficiencies of CPS, OTC, or ASS.
  Other Names: Sodium Phenylbutyrate; NaPBA

SUMMARY:
The purpose of this study is to determine whether HPN-100 is safe and tolerable in subjects with Urea Cycle Disorders.

DETAILED DESCRIPTION:
When protein is broken down in the body, nitrogen is formed. In healthy individuals, the body combines this nitrogen with other molecules to create a harmless substance called urea, which is excreted in the urine. Patients with Urea Cycle Disorders (UCD) are unable to create as much urea from nitrogen, and therefore, toxic levels of nitrogen can accumulate in the body, causing harm. To treat these patients, doctors usually have the patient consume less protein and supplement certain amino acids that may be lacking. A drug called Buphenyl® is sometimes prescribed as an adjunctive treatment for the chronic maintenance of UCD patients in order to keep ammonia levels down. Some issues with Buphenyl® include a high pill burden (up to 40 pills per day), bad taste and odor, and high sodium content. Like Buphenyl®, HPN-100 provides an alternate way for the body to dispose of nitrogen, other than through the urea cycle. Unlike Buphenyl®, HPN-100 is an odorless, tasteless, concentrated oil that does not contain large amounts of sodium.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at least 18 years old
* Signed written informed consent by patient or patient's representative
* Diagnosis of urea cycle enzyme deficiency confirmed via enzymatic or genetic testing
* Currently treated with Buphenyl® TID for a minimum of 2 weeks prior to Visit 1
* Able to perform study activities (including the ability to collect all urine in the clinic, i.e., no patients in diapers)
* Negative pregnancy test for all females of childbearing potential. All females of childbearing potential must agree to use an acceptable method of contraception throughout the study

Exclusion Criteria:

* Use of any investigational drug within 30 days of Buphenyl® Visit 1
* Active infection (viral or bacterial) or any other condition that may increase ammonia levels
* Laboratory values outside the normal range that are determined to be clinically significant by the investigator
* Any clinical or laboratory abnormality of Grade 3 or greater severity according to the Common Terminology Criteria for Adverse Events v3.0 (CTCAE) (or for conditions not covered by the CTCAE, a severe or life-threatening toxicity); except that Grade 3 elevations in liver enzymes are allowed in an otherwise clinically stable patient
* Use of any medication known to significantly affect renal clearance (e.g., probenecid) or to increase protein catabolism (e.g., corticosteroids), or other medication (e.g., valproate) known to increase ammonia levels, within the 24 hours prior to Visit 1
* Preexisting QTc interval prolongation (> 450 msec for males or > 460 msec for females)
* Other severe chronic medical conditions
* Known hypersensitivity to PAA, PBA, or benzoate
* Creatinine levels equal to or greater than 1.5 × ULN
* Liver transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Shih VE. Alternative-pathway therapy for hyperammonemia. N Engl J Med. 2007 May 31;356(22):2321-2. doi: 10.1056/NEJMe078075. No abstract available. PMID 17538092
- [Background] Enns GM, Berry SA, Berry GT, Rhead WJ, Brusilow SW, Hamosh A. Survival after treatment with phenylacetate and benzoate for urea-cycle disorders. N Engl J Med. 2007 May 31;356(22):2282-92. doi: 10.1056/NEJMoa066596. PMID 17538087
- [Derived] Mokhtarani M, Diaz GA, Rhead W, Berry SA, Lichter-Konecki U, Feigenbaum A, Schulze A, Longo N, Bartley J, Berquist W, Gallagher R, Smith W, McCandless SE, Harding C, Rockey DC, Vierling JM, Mantry P, Ghabril M, Brown RS Jr, Dickinson K, Moors T, Norris C, Coakley D, Milikien DA, Nagamani SC, Lemons C, Lee B, Scharschmidt BF. Elevated phenylacetic acid levels do not correlate with adverse events in patients with urea cycle disorders or hepatic encephalopathy and can be predicted based on the plasma PAA to PAGN ratio. Mol Genet Metab. 2013 Dec;110(4):446-53. doi: 10.1016/j.ymgme.2013.09.017. Epub 2013 Oct 8. PMID 24144944
- [Derived] Diaz GA, Krivitzky LS, Mokhtarani M, Rhead W, Bartley J, Feigenbaum A, Longo N, Berquist W, Berry SA, Gallagher R, Lichter-Konecki U, Bartholomew D, Harding CO, Cederbaum S, McCandless SE, Smith W, Vockley G, Bart SA, Korson MS, Kronn D, Zori R, Merritt JL 2nd, C S Nagamani S, Mauney J, Lemons C, Dickinson K, Moors TL, Coakley DF, Scharschmidt BF, Lee B. Ammonia control and neurocognitive outcome among urea cycle disorder patients treated with glycerol phenylbutyrate. Hepatology. 2013 Jun;57(6):2171-9. doi: 10.1002/hep.26058. Epub 2013 Jan 3. PMID 22961727

RESULTS

PARTICIPANT FLOW:
Groups:
- Buphenyl to HPN-100: HPN-100 : Subjects took prescribed dose of Buphenyl® TID (not to exceed 20g/day) at least two weeks prior to enrollment. Subjects took prescribed dose of Buphenyl® TID for first week of study, and then switched over to HPN-100 TID during a dose-escalation phase. The dose of HPN-100 was increased and the dose of Buphenyl® was decreased each week by 50 mg/kg until entire daily dose of phenylbutyrate was HPN-100. Target HPN-100 dose contained the same amount of phenylbutyrate as the subject's prescribed daily dose of Buphenyl®. Subject took HPN-100 alone for one week and then switched back to previous dose of Buphenyl for the last week of the study.
Period: Overall Study
Arm/Group | Buphenyl to HPN-100
Started | 14
Completed | 10
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Buphenyl to HPN-100: HPN-100 : Subjects will be taking prescribed dose of Buphenyl® TID (not to exceed 20g/day) at least two weeks prior to enrollment. Subjects will take prescribed dose of Buphenyl® TID for first week of study, and then switch over to HPN-100 TID during a dose-escalation phase. The dose of HPN-100 will be increased and the dose of Buphenyl® will be decreased each week by 50 mg/kg until entire daily dose of phenylbutyrate is HPN-100. Target HPN-100 dose will contain the same amount of phenylbutyrate as the subject's prescribed daily dose of Buphenyl®. Subject will take HPN-100 alone for one week and then switch back to previous dose of Buphenyl for the last week of the study.
Arm/Group | Buphenyl to HPN-100
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Secondary Outcome: Pharmacokinetics (Plasma and Urine PK Parameters of Study Drugs and Their Metabolites)
Description: measured AUC0-24 (Area under the curve from time 0 (pre-dose) to 24 hours) for each metabolite in plasma. Data were collected at 30 minutes and 1, 2, 4, 5, 6, 8, 10, 12, and 24 hours post-first dose.
Time Frame: At steady state (1 week) on each medication (Buphenyl® alone, HPN-100 alone)
Measure: Mean (Standard Deviation); unit: μg*h/mL
Units Other Than Participants: plasma
Groups:
- NaPBA Steady State: Subjects were on NaPBA TID treatment for at least 2 weeks prior to enrollment, and were thus expected to be at steady-state levels prior to enrollment. After enrollment, subjects received 1 week of NaPBA treatment before switching over to HPN-100 dose escalation phase.
- HPN-100 Steady State: After dose escalation to full dose of HPN-100 was completed, subjects received only HPN-100 for 1 week (and achieved steady state) prior to switching back to their original NaPBA treatment.
Arm/Group | NaPBA Steady State | HPN-100 Steady State
Number analyzed (Participants) | 10 | 10
Number analyzed (plasma) | 86 | 82
μg*h/mL
  AUC0-24 PBA (phenylbutyrate) in plasma | 740 (363) | 540 (325)
  AUC0-24 PAA (phenylacetate) in plasma | 596 (738) | 575 (970)
  AUC0-24 PAGN (phenylacetylglutamine) in plasma | 1133 (352) | 1098 (485)

2. Primary Outcome: Venous Ammonia Levels at the Peak and Mean TNUAC Time-normalized Area Under the Curve)
Description: Data were collected at pre-first dose and at 30 minutes and 1, 2, 4, 5, 6, 8, 10, 12, and 24 hours post first dose.
Time Frame: At steady state (1 week) on each medication (Buphenyl® alone, HPN-100 alone), and at steady state (1 week) after each dose escalation
Measure: Mean (Standard Deviation); unit: μmol/L
Units Other Than Participants: concentration of ammonia
Arm/Group | NaPBA Steady State | HPN-100 Steady State
Number analyzed (Participants) | 10 | 10
Number analyzed (concentration of ammonia) | 10 | 10
μmol/L
  in peak | 79.1 (40.1) | 56.3 (27.9)
  in TNAUC (time-normalized area under the curve) | 38.4 (19.6) | 26.5 (10.7)

3. Secondary Outcome: Drug Preference for HPN-100 or Buphenyl® (as Assessed by Global Preference Question)
Time Frame: End of Study
Measure: Number; unit: participants
Arm/Group | Buphenyl to HPN-100
Number analyzed (Participants) | 10
participants
  prefer Buphenyl | 1
  prefer HPN-100 | 9

4. Primary Outcome: Number of Subjects Experienced Adverse Events
Time Frame: during the period on 100% Buphenyl (up to 4 weeks) or HPN-100 (up to 10 weeks)
Measure: Number; unit: participants
Groups:
- Buphenyl: Subjects took prescribed dose of Buphenyl® TID (not to exceed 20g/day) at least two weeks prior to enrollment. Subjects took prescribed dose of Buphenyl® TID for first week of study before blood sample collection.
- HPN-100: HPN-100 dose contained the same amount of phenylbutyrates as the subject's prescribed daily dose of Buphenyl®. Subject took HPN-100 alone for one week to reach steady state before blood sample collection.
Arm/Group | Buphenyl | HPN-100
Number analyzed (Participants) | 14 | 10
participants | 7 | 5

5. Primary Outcome: Number of Subjects Experienced Serious Adverse Events
Time Frame: during the period subjects on 100% Buphenyl (up to 4 weeks) or HPN-100 (up to 10 weeks)
Measure: Number; unit: participants
Groups:
- HPN-100: HPN-100 dose contained the same amount of phenylbutyrate as the subject's prescribed daily dose of Buphenyl®. Subject took HPN-100 alone for one week to reach steady state before blood sample collection.
Arm/Group | Buphenyl | HPN-100
Number analyzed (Participants) | 14 | 10
participants | 1 | 0

ADVERSE EVENTS:
Description: The occurrence of adverse events was assessed by investigator assessment, clinical laboratory measurements, ECG, vitals signs measurements and symptom survey.
Groups:
- Buphenyl; HPN-100: HPN-100 : Subjects will be taking prescribed dose of Buphenyl® TID (not to exceed 20g/day) at least two weeks prior to enrollment. Subjects will take prescribed dose of Buphenyl® TID for first week of study, and then switch over to HPN-100 TID during a dose-escalation phase. The dose of HPN-100 will be increased and the dose of Buphenyl® will be decreased each week by 50 mg/kg until entire daily dose of phenylbutyrate is HPN-100. Target HPN-100 dose will contain the same amount of phenylbutyrate as the subject's prescribed daily dose of Buphenyl®. Subject will take HPN-100 alone for one week and then switch back to previous dose of Buphenyl for the last week of the study.
Arm/Group | Buphenyl | HPN-100
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/10
Other Adverse Events (participants affected / at risk) | 7/14 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buphenyl (N=14) | HPN-100 (N=10)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Buphenyl (N=14) | HPN-100 (N=10)
Nausea (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Increased Appetite (Metabolism and nutrition disorders) | 1 | 3
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Skin Odour Abnormal (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days